CLINICAL TRIAL: NCT02863120
Title: Patient Outcomes With Periarticular Liposomal Bupivacaine Injection vs Adductor Canal Block After Primary Total Knee Arthroplasty
Brief Title: Liposomal Bupivacaine vs Adductor Canal Block in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Orthopaedics, Sports and Rehabilitation Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-EXP-160402
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Knee Osteoarthritis
Keywords: Bupivacaine; Osteoarthritis; Arthritis; Joint Diseases; Ropivacaine; Anesthetics, Local; Anesthetics
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis; Joint Diseases | interventions — Bupivacaine; Ropivacaine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal bupivacaine (Active Comparator): Periarticular infiltration of 20cc of liposomal bupivacaine with 10cc of normal saline and 30cc of bupivacaine HCl administered prior to cementation of knee implants
  Interventions: Drug: liposomal bupivacaine; Drug: bupivacaine HCl; Drug: Saline
- Adductor canal and tibial nerve block (Active Comparator): Preoperative tibial nerve block with 15cc bupivacaine HCl and adductor canal block with 20cc adductor canal block. Postoperative continuous adductor canal block with 550cc ropivacaine at 8cc per hour
  Interventions: Drug: bupivacaine HCl; Drug: Ropivacaine

INTERVENTIONS:
Drug: liposomal bupivacaine
  Other Names: Exparel
  Arms: Liposomal bupivacaine
Drug: bupivacaine HCl
  Other Names: Marcaine
Drug: Ropivacaine
  Other Names: Naropin
  Arms: Adductor canal and tibial nerve block
Drug: Saline
  Arms: Liposomal bupivacaine

SUMMARY:
This study is being done to evaluate the outcomes of patients undergoing total knee replacement with two different methods of local pain control:shots of liposomal bupivacaine, a long acting anesthetic, directly into the knee during surgery or anesthetic delivered continuously to the adductor canal to provide long term pain relief. The goal is to try to find a standard protocol that provides the greatest pain relief for patients undergoing total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female between the ages of 18-65
* Patients willing and able to sign the informed consent
* Patients able to comply with follow-up requirements including self-evaluations
* Patients requiring a primary total knee replacement
* Patients with a diagnosis of osteoarthritis, traumatic arthritis, or avascular necrosis

Exclusion Criteria:

* Revision total knee arthroplasty
* Bilateral total knee arthroplasty
* Patients with inflammatory arthritis
* Patients with a body mass index (BMI) > 40
* Allergy to ropivacaine, bupivacaine, or other local anesthetic agents
* Current use of opioid drugs
* Patients with a history of total or unicompartmental reconstruction of the affected joint
* Patients that have had a high tibial osteotomy or femoral osteotomy
* Patients with neuromuscular or neurosensory deficiency, which would limit the ability to assess pain levels
* Patients with a systemic or metabolic disorder leading to progressive bone deterioration
* Patients that are immunologically compromised, or receiving chronic steroids (>30 days), excluding inhalers
* Patients' bone stock is compromised by disease or infection, which cannot provide adequate support and/or fixation to the prosthesis
* Patients with knee fusion to the affected joint
* Patients with an active or suspected latent infection in or about the knee joint
* Patients that are prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Length of stay (LOS, in days) | Participants will be followed for the duration of their hospital stay, an expected average of 1.5 days
Time to ambulation (in hours) | 2-6 hours

SECONDARY OUTCOMES:
Pain as assessed by visual analog scale (VAS) on postoperative day 0 | 6 hours
  Pain levels will be determined on postoperative day 0, 1, 2, 3, 4, and 5
Pain as assessed by visual analog scale (VAS) on postoperative day 1 | 24 hours
  Pain levels will be determined on postoperative day 0, 1, 2, 3, 4, and 5
Pain as assessed by visual analog scale (VAS) on postoperative day 2 | 48 hours
  Pain levels will be determined on postoperative day 0, 1, 2, 3, 4, and 5
Pain as assessed by visual analog scale (VAS) on postoperative day 3 | 72 hours
  Pain levels will be determined on postoperative day 0, 1, 2, 3, 4, and 5
Pain as assessed by visual analog scale (VAS) on postoperative day 4 | 96 hours
  Pain levels will be determined on postoperative day 0, 1, 2, 3, 4, and 5
Pain as assessed by visual analog scale (VAS) on postoperative day 5 | 120 hours
  Pain levels will be determined on postoperative day 0, 1, 2, 3, 4, and 5
Opioid consumption in oral morphine equivalents (OMEs, in milligrams) | Participants will be followed for the duration of their hospital stay, an expected average of 1.5 days.
Postoperative complications and adverse events | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tyler D Goldberg, MD, Principal Investigator — Texas Orthopedics
Locations (1):
- Texas Orthopedics, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No